CLINICAL TRIAL: NCT00392106
Title: Study of Focused Circumferential UltraSound for the Treatment of Atrial Fibrillation
Brief Title: High Intensity Focused Ultrasound (HIFU) Ablation System Study
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: voluntarily by Sponsor to investigate an anticipated SAE
Sponsor: ProRhythm, Inc. (Industry)
Responsible Party: Reinhard Warnking, President and CEO, ProRhythm, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-003; NCT00392106
Record Dates: First submitted 2006-10-24; First posted 2006-10-25 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; arrhythmia; AF ablation; antiarrhythmic agent; catheter ablation; pulmonary veins
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac | interventions — Propafenone; Flecainide; dofetilide; Sotalol; Amiodarone

ARMS (2):
- Control (Active Comparator): Class I or III anti-arrhythmic drug for the treatment of AF
  Interventions: Drug: propafenone; Drug: flecainide; Drug: dofetilide; Drug: sotolol; Drug: Amiodarone
- Treatment (Experimental): Pulmonary vein ablation with HIFU
  Interventions: Device: Pulmonary vein ablation

INTERVENTIONS:
Drug: propafenone — Anti-arrhythmic drug prescribed for treatment of atrial fibrillation
  Other Names: Rhyhmol
  Arms: Control
Drug: flecainide — Anti-arrhythmic drug prescribed for the treatment of Atrial fibrillation
  Other Names: Tambocor
  Arms: Control
Drug: dofetilide — Anti-arrhythmic drug prescribed for treatment of atrial fibrillation
  Other Names: Tikosyn
  Arms: Control
Drug: sotolol — Anti-arrhythmic Drug prescribed for treatment of Atrial Fibrillation
  Other Names: Betapace
  Arms: Control
Device: Pulmonary vein ablation — Electrical isolation of pulmonary vein with high-intensity focused ultrasound
  Other Names: Left atrial ablation
  Arms: Treatment
Drug: Amiodarone — Anti-arrhythmic Drug prescribed for the treatment of Atrial Fibrillation
  Other Names: Pacerone
  Arms: Control

SUMMARY:
The purpose of this study is to determine if the HIFU Pulmonary Vein Ablation System is effective in the treatment of paroxysmal Atrial Fibrillation compared to the control of best medical therapy with FDA approved antiarrhythmic drugs.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common sustained cardiac arrhythmia affecting an estimated 2.2 million persons in the United States (US). In addition to being debilitating, AF has been identified as a leading risk factor for stroke. AF is often associated with structural heart disease, but a substantial number of AF patients have little or no detectable structural heart disease. A patient with AF is up to 5 times more likely to have a stroke than the general population.

Recently, it has been demonstrated that for a significant portion of AF patients (80% - 95 %) the arrhythmia originates in one of the four pulmonary veins (PV's). Furthermore, it has been shown that isolation of this arrhythmia by ablation can, in the majority of patients (50-70%), eliminate or markedly reduce episodes of AF. Currently, there are a number of modalities being investigated to treat AF. They include radiofrequency, laser, thermal, cryo, microwave, and ultrasound ablation of targeted areas in the atrium and/or PVs.

Comparison(s): Clinical success of High Intensity Focused Ultrasound (HIFU) Ablation for Pulmonary Vein Isolation in the treatment of Atrial Fibrillation, compared to medical therapy with anti-arrhythmic drugs (AADs).

ELIGIBILITY:
Inclusion Criteria:

* Documented atrial fibrillation
* Failed or intolerant to at least 1 anti-arrhythmic drug
* Able to take anti-coagulant therapy
* Able to complete screening tests required for inclusion/exclusion criteria
* Able to take at least 1 approved anti-arrhythmic drug
* Not pregnant
* Available for follow-up for at least 12 months

Exclusion Criteria:

* Persistent or permanent atrial fibrillation
* Mitral disease
* Prior surgical treatment for atrial fibrillation
* Ablation for treatment of atrial fibrillation within 6 months
* Severe left ventricular hypertrophy
* Known untreated coagulopathy
* Unstable angina
* Prior stroke
* Uncontrolled heart failure
* Secondary causes of atrial fibrillation
* Uncorrected hyperthyroidism within 12 months
* Pulmonary embolism within 6 months
* Pneumonia or acute pulmonary disease within 3 months
* Pacemaker/ICD
* High risk for esophageal disease
* Currently enrolled in investigational drug or device study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2006-04; Primary Completion 2010-12 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Acute treatment with elimination of AF episodes | 12 months
Death, stroke, and hospitalization for recurrence of AF | within 12 months of treatment

SECONDARY OUTCOMES:
Acute treatment success | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Warren Jackman, MD, Principal Investigator — Oklahoma University Health Sciences Center; Hugh Calkins, MD, Principal Investigator — Johns Hopkins Medical Center
Locations (21):
- United States (20):
  - Fullerton Vascular Medical Group, Fullerton, California
  - University of California, Los Angeles, Los Angeles, California
  - Piedmont Hospital, Atlanta, Georgia
  - Lexington Central Baptist Hospital, Lexington, Kentucky
  - Johns Hopkins Hopsital, Baltimore, Maryland
  - Lahey Clinic, Burlington, Massachusetts
  - Beaumont Hospital, Royal Oak, Michigan
  - New York University Hospital, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Wake Forest University Health Systems, Winston-Salem, North Carolina
  - Hillcrest Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University Heart Center, Columbus, Ohio
  - Oklahoma University Health Sciences Center, Oklahoma City, Oklahoma
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Cardiac Arrhythmia Research, Austin, Texas
  - University of Texas, Southwestern, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
- Homolka Hospital, Prague, Czechia